CLINICAL TRIAL: NCT03403257
Title: Brain Attack Surveillance in Corpus Christi--Cognitive (BASIC-Cognitive)
Acronym: BASIC-C
Status: Active, not recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Lewis Morgenstern, Professor, University of Michigan
Other Study IDs: R01NS100687 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Dementia Alzheimers; Dementia, Vascular; Dementia, Mixed
Keywords: Caregiving; Hispanic; Mexican American; Epidemiology; Community
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Mixed Dementias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Subjects with cognitive impairment: Subjects with MoCA <26
  Interventions: Other: No interventions
- Caregivers: Primary caregivers of subjects
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No intervention

SUMMARY:
The Mexican American population in the U.S. is rapidly growing and aging. This project seeks to determine the prevalence and outcomes of cognitive impairment and dementia in Mexican Americans. It also seeks solutions to help patients with cognitive impairment and dementia and their caregivers get the resources they need.

DETAILED DESCRIPTION:
Hispanic/Latinos will comprise more than 30% of the U.S. population by mid-century, and Mexican Americans account for the largest share of this growing segment of society. This proposal aims to use door-to-door surveillance in Nueces County, Texas, a non-immigrant, bi-ethnic community, to determine the prevalence and trajectory over time of cognitive impairment and dementia in Mexican Americans and non Hispanic whites. The study will elucidate the mechanisms that explain the hypothesized ethnic disparity in Alzheimer's disease and Alzheimer-related dementias by evaluating the roles of vascular disease risk factors, educational attainment and socio-economic status among others. This research will also delve deeply into the differences in informal caregiving for Mexican American and non Hispanic whites with cognitive impairment and dementia. Caregiver burden and mental and physical health of caregivers will be examined toward efforts to develop interventions that build resilience in caregivers. A novel ability of this population-based study is to examine community resources for both patients and caregivers, and how these provisions differ by ethnicity. Using a rigorous mixed methods approach the study will identify the gap between available resources and needs for those with cognitive impairment and dementia. In this way we will be well positioned to propose ethnic-specific testable interventions that promote mental and physical health for those with cognitive impairment and dementia, as well as for those family members who provide the care. This research will therefore lead to improved well-being, autonomy and outcomes among those with cognitive impairment and dementia and their caregivers. The investigative team members have conducted research in this community for 20 years and are experts in Mexican American culture and health, cognitive impairment and dementia, epidemiologic methods, community needs assessment and health behavior research. As the Mexican American population continues its tremendous growth and aging it is vitally important to better understand the prevalence and outcomes of cognitive impairment and dementia in this population, and to rapidly develop interventions that address the burden of these common conditions in Mexican American adults, families, and communities.

ELIGIBILITY:
Inclusion Criteria:

1. >64 years of age
2. MoCA < 26
3. Nueces County resident at least 6 months a year
4. English or Spanish speaking
5. Community dwelling or nursing home

Exclusion Criteria: none

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Self-described
Study Population: Residents of Nueces County, Texas
Sampling Method: Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mild cognitive impairment and dementia in Mexican Americans and non Hispanic whites | 2 year data collection
  Prevalence estimates
Trajectory of cognitive function in Mexican Americans and non Hispanic whites | 2 year follow-up after baseline
  Change in cognitive function among subjects entered at baseline
Caregiver outcomes and changes over time | 4 years
  Comparative caregiver outcomes among Mexican Americans and non Hispanic whites

SECONDARY OUTCOMES:
Needs and community available resources for cognitive impairment | 2 years
  An asset map and determination of needs

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Morgenstern, MD, Principal Investigator — University of Michigan
Locations (1):
- Corpus Christi Nueces County Health District, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing plan conforms to NIH rules.

REFERENCES:
- [Background] Briceno EM, Mehdipanah R, Gonzales X, Heeringa S, Levine DA, Langa KM, Garcia N, Longoria R, Morgenstern LB. Methods and Early Recruitment of a Community-Based Study of Cognitive Impairment Among Mexican Americans and Non-Hispanic Whites: The BASIC-Cognitive Study. J Alzheimers Dis. 2020;73(1):185-196. doi: 10.3233/JAD-190761. PMID 31771059
- [Background] Briceno EM, Mehdipanah R, Gonzales XF, Heeringa SG, Levine DA, Langa KM, Zahs D, Garcia N, Longoria R, Morgenstern LB. Bilingualism, assessment language, and the Montreal Cognitive Assessment in Mexican Americans. J Am Geriatr Soc. 2021 Jul;69(7):1971-1981. doi: 10.1111/jgs.17209. Epub 2021 May 7. PMID 33963535
- [Background] Mehdipanah R, Briceno EM, Gonzales XF, Heeringa SG, Levine DA, Langa KM, Garcia N, Longoria R, Morgenstern LB. Dementia care needs for individuals and caregivers among Mexican Americans and non-Hispanic Whites. Aging Ment Health. 2022 Aug;26(8):1630-1641. doi: 10.1080/13607863.2021.1925222. Epub 2021 Jun 7. PMID 34096422
- [Background] Briceno EM, Mehdipanah R, Gonzales XF, Heeringa SG, Levine DA, Langa KM, Zahs D, Garcia N, Longoria R, Vargas A, Morgenstern LB. Differential Relationships Between the Montreal Cognitive Assessment and Informant-Rated Cognitive Decline Among Mexican Americans and Non-Hispanic Whites. J Geriatr Psychiatry Neurol. 2022 Jul;35(4):555-564. doi: 10.1177/08919887211029383. Epub 2021 Jul 22. PMID 34291678
- [Background] Khan N, Garcia N, Mehdipanah R, Briceno EM, Heeringa SG, Levine DA, Gonzales XF, Langa KM, Longoria R, Morgenstern LB. Lack of Any Caregiving for Those with Dementia. J Alzheimers Dis. 2022;86(2):531-535. doi: 10.3233/JAD-215418. PMID 35068465
- [Background] Gonzales XF, Heeringa SG, Briceno EM, Mehdipanah R, Levine DA, Langa KM, Garcia N, Longoria R, Morgenstern LB. Mexican Americans Participate in Research More than Expected while non-Hispanic Whites Participate Less than Expected. J Health Care Poor Underserved. 2022;33(2):590-596. doi: 10.1353/hpu.2022.0049. PMID 35574862
- [Background] Mehdipanah R, Briceno EM, Heeringa SG, Gonzales XF, Levine DA, Langa KM, Garcia N, Longoria R, Chang W, Morgenstern LB. Neighborhood SES and Cognitive Function Among Hispanic/Latinx Residents: Why Where You Live Matters. Am J Prev Med. 2022 Oct;63(4):574-581. doi: 10.1016/j.amepre.2022.04.016. Epub 2022 Jun 9. PMID 35691843
- [Background] Becker CJ, Heeringa SG, Chang W, Briceno EM, Mehdipanah R, Levine DA, Langa KM, Gonzales XF, Garcia N, Longoria R, Springer MV, Zahuranec DB, Morgenstern LB. Differential Impact of Stroke on Cognitive Impairment in Mexican Americans and Non-Hispanic White Americans. Stroke. 2022 Nov;53(11):3394-3400. doi: 10.1161/STROKEAHA.122.039533. Epub 2022 Aug 12. PMID 35959679
- [Derived] Martins-Caulfield J, Mehdipanah R, Briceno EM, Chang W, Heeringa SG, Gonzales XF, Levine DA, Langa KM, Zahuranec DB, Garcia N, Morgenstern LB. Dementia Diagnosis Unawareness and Caregiver Burden in a Multi-ethnic Cohort. J Gen Intern Med. 2025 Jul;40(10):2284-2291. doi: 10.1007/s11606-024-09333-1. Epub 2025 Jan 14. PMID 39808391
- [Derived] Morgenstern LB, Briceno EM, Mehdipanah R, Chang W, Lewandowski-Romps L, Gonzales XF, Levine DA, Langa KM, Garcia N, Khan N, Zahuranec DB, Heeringa SG. A Community-Based Study of Dementia in Mexican American and Non-Hispanic White Individuals. J Alzheimers Dis. 2024;97(2):649-658. doi: 10.3233/JAD-230729. PMID 38143352
- [Derived] Khan N, Briceno EM, Mehdipanah R, Lewandowski-Romps L, Heeringa SG, Garcia N, Levine DA, Langa KM, Morgenstern LB. A community-based study of reporting demographic and clinical information concordance between informants and cognitively impaired participants. Aging Clin Exp Res. 2023 Jul;35(7):1571-1576. doi: 10.1007/s40520-023-02435-6. Epub 2023 May 19. PMID 37204754